CLINICAL TRIAL: NCT02765308
Title: The Contribution of Altered Aqueous Dynamics in the Development of Raised Intraocular Pressure in Patients With Uveitis
Brief Title: Aqueous Humor Dynamics and Hypertensive Uveitis
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 136787
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Uveitic Glaucoma; Anterior Uveitis
Keywords: Uveitis; Glaucoma; Aqueous humor dynamics
MeSH Terms: conditions — Uveitis, Anterior; Uveitis; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy volunteers: healthy age matched with cases volunteers as controls
- Uveitis with raised IOP: Recurrent (> 5 attacks) idiopathic acute anterior uveitic with raised intraocular pressure
- Uveitis with with normal IOP: Recurrent (> 5 attacks) idiopathic acute anterior uveitic with normal intraocular pressure

SUMMARY:
Uveitis is a disease that affects over 2 million people around the globe, and can ultimately lead to blindness. The proportion of patients with uveitis who become blind has not been reduced over the past 30 years, and this is therefore an area that demands further research. One of the major causes of blindness in uveitic patients is the development of uveitic glaucoma, which occurs in 10-20% of uveitic eyes. This is likely to occur for reasons related to the uveitis itself, but can also be caused as a side effect of the corticosteroids used to treat uveitis. The raised IOP in uveitis is more difficult to treat than other types of glaucoma.

To enable more effective treatment of uveitic glaucoma, the investigators need to understand more clearly the mechanisms which underlie this process. The investigators therefore propose a study to examine the contribution of altered aqueous dynamics to the development of raised IOP in uveitis.

DETAILED DESCRIPTION:
The investigators propose to undertake a cross-sectional observational study of patients with recurrent idiopathic acute anterior uveitis, to determine the relative contributions of altered aqueous production and drainage to the development of raised IOP in these patients.

Methods

Study Design A cross sectional observational study

Patient Selection All subjects attending the uveitis and glaucoma clinics at St Thomas' Hospital will be eligible to be included in the study if they fulfil the inclusion/exclusion criteria as below.

30 patients will be included from each of these three group of patients: 1) recurrent (> 5 attacks) idiopathic acute anterior uveitic with raised intraocular pressure; 2) recurrent (> 5 attacks) idiopathic acute anterior uveitic without raised intraocular pressure; 3) healthy age matched volunteers as controls. Patients on glaucoma treatment will be washed out for one month before measurement.

Examination Schedule and Methods

1. Visual acuity:

   Visual acuity is measured before pupil dilation, tonometry, gonioscopy, or any other technique that could affect vision. Two different techniques are used to measure visual acuity, including Snellen and ETDRS visual acuity testing. Refraction is performed prior to formal measurement of visual acuity by either technique.

   Subjective Refraction:

   It is permissible to use a phoropter or trial frame to determine best-corrected Snellen visual acuity. The left eye is occluded first. An approximate beginning refraction may be determined by retinoscopy, automated refraction, or a subjective refraction from a prior visit. The sphere is refined first. The cylinder is then refined, first the axis followed by the power. Finally, the sphere is rechecked. The right eye is then occluded, and the procedure is repeated for the left eye.

   If the patient wears contact lenses and has glasses also, he or she is instructed not to wear the contact lenses on the day of the assessment. Patients unwilling to discontinue contact lens use after surgery will be excluded from the study. In the event that the patient either has no glasses or has forgotten the instructions and reported for the assessment wearing contact lenses, the contact lenses are removed and at least thirty minutes allowed to elapse before subjective refraction and visual acuity testing is performed.

   ETDRS Visual Acuity:

   The logmar visual acuity testing for the Uveitic Glaucoma study has been adapted from the Early Treatment of Diabetic Retinopathy (ETDRS) at 4 metres. The logmar visual acuity scale facilitates statistical analysis and simplifies quantification of acuity at various distances. The right eye is tested with ETDRS logmar chart 1, then the left eye is tested with ETDRS logmar chart 2. Each chart is hidden from view until the eye being examined is ready for testing.

   Snellen Visual Acuity:

   Snellen visual acuity may be measured using any standard visual acuity chart. The same type of chart must be used throughout the duration of the study. Standardized refraction is performed prior to Snellen visual acuity testing.
2. Slit lamp biomicroscopy Examination of the anterior segment using slit lamp biomicroscopy will be performed. Slit lamp biomicroscopy may be performed with any commercially available instrument, and it is used in a standard fashion starting anteriorly and working posteriorly.
3. Gonioscopy Gonioscopy is performed with the patient sitting at the slit lamp using either a Zeiss type four-mirror gonioprism or Goldmann single- or three-mirror lens.
4. Pachymetry Central corneal thickness is measured with ultrasound pachymetry. The right eye is tested first. A drop of 0.5% proparacaine is instilled for anesthesia. The patient is asked to look straight ahead at a distant object or fixation target. The pachymeter probe is lined up with the center of the pupil and slowly advanced until it contacts the cornea. The probe is withdrawn when an audible signal is made indicating that a measurement has been recorded. The patient is instructed to blink. The procedure is repeated to obtain three separate readings, and the investigator records the measurements. After testing of the right eye is complete, the same technique is applied to testing of the left eye.
5. Biometry A Carl Zeiss IOL Master will be used to carry out biometry and assess anterior chamber depth using A-scan ultrasound. This is a non-contact examination technique.
6. Fundoscopy A dilated fundus examination is performed. After pupil dilation with appropriate mydriatics, the optic nerve and posterior pole are examined at the slit lamp using Volk 90 diopter, 78 diopter, or 60 diopter lens.
7. Flurophotometry The night before (10 PM) the fluorophotometric scans, participants will self-administered 3 to 6 drops of fluorescein sodium 2% (Minims, Bausch&Lomb, UK) topically into both eyes at 5 minutes interval depending on their age (age 25 years or younger, 5-6 drops; age 26 to 35 years, four drops; over 35 years of age, three drops). Fluorophotometry will be performed in both eyes using a scanning ocular fluorophotometer from 9AM to 12PM (FM-2, Fluorotron Master Ocular Fluorophotometer; OcuMetrics, Mountain View, California). The aqueous turnover protocol will be used to calculate the aqueous flow rate. Duplicate or triplicate scans will be collected and repeated at 1 hour intervals for 4 measurements to determine the aqueous flow rate (Ft). Following each set of scans, IOP will be measured using pneumatonometry (Model 30 Classic, Reichert Ophthalmic Instruments, Depew, New York). IOP will be recorded as the arithmetic mean of a total of 12 measurements per eye: 3 measurements every hour alternating between eyes.
8. Tonography Tonographic outflow facility (C) will be performed using an electronic Schiøtz tonographer (Model 720, Berkeley Bioengineering Inc, USA) at 10AM. The facility of outflow will be calculated from the rate of decay of intraocular pressure in the supine position during application of a recording Schiøtz tonometer over a period of 4 minutes with a standard 5.5 gram weight. The "R" values of the curve at every 30-second time point will be manually entered into the McLaren tonography computer program. The program fits a second-degree polynomial by least squares to the nine data points and determines the best-fit values for time 0 and time 4 minutes by extrapolation.

   Uveoscleral outflow will be calculated using the Goldmann's equation with an assumed episcleral venous of 8, 9, 10 or 11 mmHg. Ft is the rate of aqueous humor formation, C is the tonographic facility of outflow, IOP is the intraocular pressure, Pv is the episcleral venous pressure and Fu is the uveoscleral outflow.

   Ft = C (IOP-Pv) +Fu Fu = Ft-C (IOP-Pv)

   Only one randomly (Excel random number generator) chosen eye per participant will be included in the data analysis when both eyes fulfilled the inclusion criteria.
9. Visual fields Quantitative automated perimetry is performed using the Humphrey Field Analyzer. Visual field testing is performed before tonometry, gonioscopy, or any other technique that could affect vision. A visual field should be attempted in any eye that has sufficient vision to permit finger counting at two feet. Eyes with poor central vision may have an intact, off-center island of vision which may be measured with perimetry.

A 24-2 threshold test is performed in all patients using a size III white stimulus. Visual field testing may be performed with the Swedish Interactive Thresholding Algorithm (SITA) or full threshold strategy, but the same testing strategy must be used throughout the duration of the study. The pupil diameter should be 3 mm or greater before visual field testing is undertaken, and this may require pharmacologic dilation. Standardized refraction is performed to determine the patient's distance refraction and best-corrected visual acuity prior to visual field testing. The age appropriate plus lens is added to the distance refraction. Patient education is provided, and the instrument is set up for the test. The technician should monitor the patient during testing. Visual fields are performed preoperatively (within one month of enrollment in the study) and annually thereafter. Copies of all visual fields are faxed to the Statistical Coordinating Center for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with idiopathic recurrent anterior uveitis with or without raised IOP.
2. Normal healthy subjects with no ocular problems (other than refractive error) and IOP at screening < 21mmHg.
3. Age >18 years.
4. Adequate cognitive function and ability to understand verbal and written information in English.

Exclusion Criteria:

1. Other secondary glaucomas including pigment dispersion syndrome and pseudoexfoliation.
2. Normotensive glaucoma.
3. Primary angle closure.
4. Ocular trauma.
5. Intraocular or keratorefractive surgery.
6. Use of systemic medication that may affect aqueous humour production such as beta-blockers.
7. A history of allergy or hypersensitivity to fluorescein.
8. Any abnormalities preventing reliable IOP or fluorophotometric readings.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients will be included from each of these three group of patients: 1) recurrent (> 5 attacks) idiopathic acute anterior uveitic with raised intraocular pressure; 2) recurrent (> 5 attacks) idiopathic acute anterior uveitic without raised intraocular pressure; 3) healthy age matched volunteers as controls.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Facility of outflow | day 1 only (study completion)
  Tonographic outflow facility (C) will be performed using an electronic Schiøtz tonographer (Model 720, Berkeley Bioengineering Inc, USA) at 10AM
Rate of aqueous flow (measured by fluorophotometry). | Four times during the morning through day 1 only (study completion)
  Fluorophotometry will be performed in both eyes using a scanning ocular fluorophotometer from 9AM to 12PM (FM-2, Fluorotron Master Ocular Fluorophotometer; OcuMetrics, Mountain View, California). The aqueous turnover protocol will be used to calculate the aqueous flow rate. Duplicate or triplicate scans will be collected and repeated at 1 hour intervals for 4 measurements to determine the aqueous flow rate (Ft).

CONTACTS AND LOCATIONS:
Overall Officials: K Sheng l, MD, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Derived] Ho H, Daas A, Ho J, Alaghband P, Galvis EA, de Antonio Ramirez A, Grassi P, Lim R, Lim KS. Intraocular pressure changes following topical ocular hypotensive medications washout. Br J Ophthalmol. 2021 Feb;105(2):205-209. doi: 10.1136/bjophthalmol-2019-315778. Epub 2020 Apr 10. PMID 32277009